CLINICAL TRIAL: NCT07152769
Title: Iparomlimab and Tuvonralimab Combined With Gemcitabine and Cisplatin (GC) Versus Sintilimab Combined With GC as First-Line Treatment for Advanced Intrahepatic Cholangiocarcinoma: A Single-Center, Open-Label, Randomized Controlled Phase II Study
Brief Title: Iparomlimab and Tuvonralimab Combined With GC in Advanced ICC
Acronym: ITUS
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Lu Wang, MD, PhD, MD,PhD, Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2507325-6
Record Dates: First submitted 2025-08-26; First posted 2025-09-03 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-08

CONDITIONS: Advanced Intrahepatic Cholangiocarcinoma
Keywords: ICC; Iparomlimab and Tuvonralimab; Sintilimab
MeSH Terms: interventions — sintilimab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Iparomlimab and Tuvonralimab + GC (Experimental): Iparomlimab and Tuvonralimab combined with Gemcitabine and Cisplatin
  Interventions: Drug: Iparomlimab and Tuvonralimab + GC
- Sintilimab + GC (Active Comparator): Sintilimab cimbined with Gemcitabine and Cisplatin
  Interventions: Drug: Sintilimab + GC

INTERVENTIONS:
Drug: Iparomlimab and Tuvonralimab + GC — Iparomlimab and Tuvonralimab: 5mg/kg, iv, q3w; Gemcitabine: 1000 mg/m2，iv，d1、d8，q3w; Cisplatin: 25 mg/m2，iv，d1、d8，q3w
  Arms: Iparomlimab and Tuvonralimab + GC
Drug: Sintilimab + GC — Sintilimab: 5mg/kg, iv, q3w; Gemcitabine: 1000 mg/m2，iv，d1、d8，q3w; Cisplatin: 25 mg/m2，iv，d1、d8，q3w.
  Arms: Sintilimab + GC

SUMMARY:
This study is a randomized, controlled, open-label, single center clinical study. This study is designed to evaluate the efficacy and safety of Iparomlimab and Tuvonralimab Combined With GC versus Sintilimab Combined With GC as first-line therapy in advanced ICC.

DETAILED DESCRIPTION:
This study is a randomized, controlled, open-label, single center clinical study. This study is designed to evaluate the efficacy and safety of Iparomlimab and Tuvonralimab Combined With GC versus Sintilimab Combined With GC as first-line therapy in advanced ICC.

The primary endpoint is investigator-assessed 6-month Progression-Free Survival Rate . Secondary endpoints include ORR, DCR, DoR, TTR, PFS, OS, AE.

This study plans to enroll 104 patients with advanced ICC. These patients are assigned in a 1:1 ratio to the Iparomlimab and Tuvonralimab Combined With GC group (experimental group) and Sintilimab Combined With GC group (control group).

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent obtained prior to any trial-related procedures.
* Male or female， ≥18 years and ≤75 years.
* Histologically confirmed unresectable advanced or metastatic intrahepatic cholangiocarcinoma (ICC). Patients who developed recurrence more than 6 months after radical surgery are eligible. If adjuvant therapy (chemotherapy and/or radiotherapy) was received, recurrence must have occurred more than 6 months after completion of adjuvant therapy.
* At least one measurable tumor lesion according to RECIST version 1.1 criteria.
* No prior systemic therapy (chemotherapy, targeted therapy, or immunotherapy) for advanced/metastatic disease.
* Life expectancy of at least 12 weeks.
* ECOG Performance Status (PS) of 0 or 1.
* Subjects must meet the following laboratory parameters: 1)Absolute Neutrophil Count (ANC): ≥ 1.5 × 10⁹/L (without granulocyte colony-stimulating factor support within the last 14 days). 2)Platelets: ≥ 100 × 10⁹/L (without transfusion within the last 14 days). 3)Hemoglobin: > 9 g/dL (without transfusion or erythropoietin use within the last 14 days). 4)Total Bilirubin: ≤ 1.5 × Upper Limit of Normal (ULN). 5)Aspartate Aminotransferase (AST), Alanine Aminotransferase (ALT): ≤ 2.5 × ULN. 6)Creatinine Clearance: Calculated creatinine clearance (using the Cockcroft-Gault formula) ≥ 60 mL/min.
* The subject is willing and able to comply with the protocol during the study period, including receiving treatment, adhering to contraceptive measures, and attending scheduled visits and examinations (including follow-up).

Exclusion Criteria:

* Previous treatment with agents targeting stimulatory or co-inhibitory T-cell receptors other than PD-1/PD-L1 (e.g., CTLA-4, OX-40, CD137).
* Systemic administration of Chinese herbal medicines with claimed anti-tumor indications or immunomodulatory agents (including thymosin, interferon, interleukin; excluding local use for pleural effusion control) within 2 weeks prior to the first dose.
* History of active autoimmune disease requiring systemic therapy (e.g., disease-modifying agents, corticosteroids, or immunosuppressants) within 2 years prior to the first dose. Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement for adrenal or pituitary insufficiency) is not considered systemic therapy. Known history of primary immunodeficiency.

Subjects with only positive autoimmune antibodies must be evaluated by the Investigator to confirm the absence of an autoimmune disease.

* Current systemic corticosteroid therapy (>10 mg/day prednisone equivalent) or any other form of immunosuppressive therapy within 4 weeks prior to the first study dose.
* Presence of clinically uncontrolled pleural effusion or ascites (subjects who do not require drainage or whose effusion shows no significant increase for ≥3 days after stopping drainage may be enrolled).
* Known history of allogeneic organ transplantation (excluding corneal transplants) or allogeneic hematopoietic stem cell transplantation.
* Known hypersensitivity to the active pharmaceutical ingredients or excipients of the investigational products used in this study.
* Failure to recover adequately (i.e., to ≤ Grade 1 or baseline, excluding alopecia or fatigue) from toxicities and/or complications of any prior interventions before initiation of study treatment.
* Known history of Human Immunodeficiency Virus (HIV) infection (i.e., HIV 1/2 antibodies positive).
* Untreated active hepatitis B (defined as HBsAg positive with detectable HBV-DNA exceeding the upper limit of normal (ULN) at the central laboratory of the participating site).
* Active hepatitis C virus (HCV) infection (HCV antibody positive and HCV-RNA levels above the lower limit of detection).
* Administration of a live attenuated vaccine within 4 weeks prior to the first dose.
* Positive pregnancy test within 7 days prior to the first dose or currently breastfeeding, for women of childbearing potential.
* Presence of any severe and/or uncontrolled systemic disease/disorder.
* Any medical condition (including psychiatric or substance abuse disorders), prior/concomitant treatment, or clinically significant laboratory abnormality that, in the investigator's opinion, would:Adversely affect trial data integrity, Limit the subject's ability to complete the study, Or pose undue risk to the subject.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Estimated)
Dates: Start 2025-10-15 (Estimated); Primary Completion 2028-02-29 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
6-month progression-free survival | 6 months
  Defined as the proportion of subjects who remain free of disease progression or death within 6 months from the start of the first study treatment.

SECONDARY OUTCOMES:
Progression-Free Survival (PFS) | up to approximately 2 years.
  Defined as the time from randomization to the first documented radiological disease progression or death (whichever occurs first).
Objective Response Rate (ORR) | up to approximately 2 years.
  Defined as the proportion of subjects achieving a Complete Response (CR) or Partial Response (PR) among all subjects.
Disease Control Rate (DCR) | up to approximately 2 years.
  Defined as the proportion of subjects achieving a Complete Response (CR), Partial Response (PR), or Stable Disease (SD) among all subjects.
Duration of Response (DOR) | up to approximately 2 years.
  Defined as the time from the first documented response (CR or PR) to disease progression or death (whichever occurs first).
Time to Response (TTR) | up to approximately 2 years.
  Defined as the time from randomization to the first documented Complete Response (CR) or Partial Response (PR).
Overall Survival (OS) | up to approximately 2 years.
  Defined as the time from randomization to death from any cause.
Adverse Events | up to approximately 2 years.
  AE assessed by NCI-CTCAE v5.0.

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China